CLINICAL TRIAL: NCT02420938
Title: Urelumab (CD137 mAb) Combined With Rituximab for Relapsed, Refractory or High-risk Untreated Patients With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Brief Title: Urelumab (CD137 mAb) With Rituximab for Relapsed, Refractory or High-risk Untreated Chronic Lymphocytic Leukemia (CLL) Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0932; NCI-2015-00805 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Leukemia
Keywords: Leukemia; Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Lymphoma; SLL; Refractory/relapsed; High-risk molecular features; Rituximab; Rituxan; Urelumab
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Rituximab; urelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab + Urelumab (Experimental): Participants receive Rituximab 375 mg/m2 by vein weekly for the first 4 weeks (Days 1, 8, 15, 22) then the day prior to each subsequent dose of Urelumab for the 12-week course. Urelumab 8 mg by vein given every 3 weeks for 4 doses, starting Day 2 of the course. Urelumab doses administered approximately 24 hours after the Rituximab doses. Up to two 12-week courses of treatment administered (total of maximum 12 doses of Rituximab and 8 doses of Urelumab).
  Interventions: Drug: Rituximab; Drug: Urelumab

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 by vein weekly for the first 4 weeks (Days 1, 8, 15, 22) then the day prior to each subsequent dose of Urelumab for the 12-week course.
  Other Names: Rituxan
Drug: Urelumab — 8 mg by vein given every 3 weeks for 4 doses, starting Day 2 of the 12-week course.

SUMMARY:
The goal of this clinical research study is to learn if urelumab given in combination with rituximab can help to control CLL or SLL. The safety of the drug combination will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive rituximab by vein over 4-6 hours on Days 1, 8, 15, 22, 43, and 64 of each 84 day (12 week) cycle.

You will receive urelumab by vein over about 1 hour on Days 2, 23, 44, and 65 of each cycle.

There will be a 2-week period between each study cycle.

Study Visits:

On Days 1, 8, 15, 22, 43, and 64 of each cycle:

* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a physical exam.

On Days 2, 29, 36, 50, 57, 71, and 78 of each cycle, blood (about 2 tablespoons) will be drawn for routine tests.

At the end of each cycle (about Day 85):

* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a physical exam.
* You will have a bone marrow aspiration and biopsy to check the status of the disease.
* You will have a CT or PET scan to check the status of the disease.

You will have blood draws, CT scans (or PET scans) and/or bone marrow aspiration and biopsies at any time that the doctor thinks it is needed while you are on study.

Length of Study:

You may receive up to 2 cycles of study drugs. However, your study doctor may allow you to receive the study drugs beyond Cycle 2. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

End-of-Study Visit:

If you are taken off study for any reason, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a bone marrow aspirate and CT or PET scan to check the status of the disease.

Long-Term Follow-Up:

After you are no longer on study, 1 time every month:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.

Every 3 months, if the doctor thinks it is needed, you will have a bone marrow aspirate and CT or PET scan to check the status of the disease.

Other Testing:

The study staff may ask you to take part in other MD Anderson clinical research study (PA13-0291) for additional research testing. The study doctor will discuss this with you and, if you decide to take part, you will sign a separate consent document.

This is an investigational study. Urelumab is not FDA approved or commercially available. Rituximab is FDA approved and commercially available for the treatment of patients with CLL. The use of these drugs in combination is investigational. The study doctor can explain how the drugs are designed to work.

Up to 24 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will have a diagnosis of CLL or SLL who meet one or more criteria for active disease as defined by the International Working Group for CLL (IWCLL) and are relapsed and/or refractory after at least one prior therapy.
2. Age 18 years or older.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status </= 2.
4. Patients must have adequate renal and hepatic function: -- Serum bilirubin </= 1.5 x upper limit of normal (ULN). For patients with Gilbert's disease, serum bilirubin up to </= 3 x ULN is allowed provided normal direct bilirubin, -- Serum creatinine </= 1.5 x ULN, -- ALT and AST </= 3 x ULN.
5. Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotrophin (Beta-hCG) pregnancy test result within 24 hours prior to the first dose of treatment and must agree to use an effective contraception method during the study and for 12 months following the last dose of the study drugs. Females of non- childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy. Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 31 weeks following the last dose of study drugs. Acceptable methods of contraception are condoms with contraceptive foam; oral, implantable or injectable contraceptives; contraceptive patch; intrauterine device; diaphragm with spermicidal gel; or a sexual partner who is surgically sterilized or post-menopausal.
6. Patients or their legally authorized representative must provide written informed consent.

Exclusion Criteria:

1. Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized prostate cancer. If patients have another malignancy that was treated within the last 2 years, such patients may be enrolled if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at MD Anderson Cancer Center and after consultation with the Principal Investigator
2. Any major surgery, radiotherapy, chemotherapy, biologic therapy, immunotherapy, experimental therapy within 4 weeks prior to the first dose of the study drugs. For oral targeted therapies (such as ibrutinib, idelalisib, venetoclax), a washout of 3 days is allowed. Note: Prior treatment with anti CD20 monoclonal antibody, anti CD52 monoclonal antibody and lenalidomide are allowed. Prior treatment with anti-CTLA-4 and anti-PD1 therapies is allowed after a wash-out of 5 half-lives.
3. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, (third-degree AV block, ventricular tachycardia, atrial fibrillation with rapid ventricular rate (HR >100 bpm)),congestive heart failure, or myocardial infarction within 2 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
4. History of stroke or cerebral hemorrhage within 2 months.
5. Patients who have uncontrolled hypertension (defined as sustained systolic blood pressure >/= 160 mmHg or diastolic >/= 100 mmHg).
6. Known evidence of active cerebral/meningeal CLL. Patients may have history of CNS leukemic involvement if definitively treated with prior therapy and no evidence of active disease at the time of registration.
7. Known active, uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia requiring steroid therapy.
8. Patients with autoimmune diseases are excluded: Patients with a history of Inflammatory Bowel Disease (including Crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis, systemic lupus erythematosus, Wegener's granulomatosis).
9. Patients with previous allogeneic stem cell transplant (SCT) within 6 months or with active acute or chronic graft-versus host disease are excluded. Patients must be off immunosuppression for GVHD for at least 30 days before cycle 1 day 1.
10. Patients with organ allografts (such as renal transplant) are excluded.
11. History of any hepatitis (e.g., alcohol or non-alcohol steatohepatitis (NASH), auto immune, or grade 3-4 drug-related hepatitis).
12. Patients who are on high-dose steroids (doses >10mg/day of prednisone or equivalent) or immune suppression medications. Note: Patients on high-dose steroids (doses >10mg/day of prednisone or equivalent) or immune suppression medications are eligible provided these drugs are discontinued at least 3 days prior to starting on the study drugs.
13. Patients with uncontrolled active infection (viral, bacterial, and fungal) are not eligible.
14. Current or chronic hepatitis B or C infection, or known seropositivity for HIV. Note: Patients with previous history of Hepatitis B (who have cleared the infection and have natural immunity, i.e. Hep B core antibody positive cases) are excluded if prophylaxis against Hep B reactivation with antiviral agents (such as entecavir) is recommended, after consultation with gastroenterologist/hepatologist or infectious disease team.
15. Patient is pregnant or breast-feeding.
16. Concurrent use of investigational therapeutic agent.
17. Patients may not receive other concurrent chemotherapy, radiotherapy, or immunotherapy. Localized radiotherapy to an area not compromising bone marrow function does not apply.
18. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study.
19. Patients with Richter's transformation are not allowed in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response (OR) of Urelumab and Rituximab in Participants with High-Risk Chronic Lymphocytic Leukemia /Small Lymphocytic Lymphoma (CLL/SLL). | 12 weeks
  Response assessed by investigator, based on physical examinations, CT scans, laboratory results, and bone marrow examinations, based on modified 2008 IWCLL criteria for response for chronic lymphocytic leukemia (CLL). Overall response (OR) includes complete remission (CR), CR with incomplete marrow recovery (CRi) or partial remission (PR). Minimal residual disease (MRD) assessed in bone marrow by multi-color flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, MBBS, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org